CLINICAL TRIAL: NCT01771211
Title: Impact of Transcranial Direct Current Stimulation on Language Functions in Mild Cognitive Impairment: A Proof-of-principle Study and Neural Correlates
Brief Title: Impact of Transcranial Direct Current Stimulation on Language Functions in Mild Cognitive Impairment
Acronym: STIMCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: German Research Foundation (Other)
Responsible Party: Principal Investigator, Marcus Meinzer, Creutzfeld Fellow, Charite University, Berlin, Germany
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: FL379101
Record Dates: First submitted 2013-01-14; First posted 2013-01-18 (Estimated); Last update posted 2013-08-22 (Estimated); Status verified 2013-08

CONDITIONS: Mild Cognitive Impairment
Keywords: MCI; Word-retrieval; tDCS; fMRI
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- anodal tDCS (Experimental): anodal tDCS will be administered for 20 minutes with 1 milliampere (1 mA) to the left inferior frontal gyrus
  Interventions: Device: tDCS
- sham tDCS (Sham Comparator): sham tDCS will be administered to the left inferior frontal gyrus
  Interventions: Device: tDCS

INTERVENTIONS:
Device: tDCS — anodal tDCS will be delivered with a constant current of 1 mA during resting-state and task-related fMRI and will continue until the end of the word-generation task. For both stimulation conditions (atDCS, sham) the current will be initially increased in a ramp-like fashion over 10 s, eliciting a tingling sensation on the scalp that fades over seconds. During sham stimulation the current will be turned off after 30 s.
  Other Names: DC-Stimulator Plus, neuroConn GmbH

SUMMARY:
The purpose of this study is to determine if non-invasive electrical brain stimulation can improve word-retrieval in Mild Cognitive Impairment (MCI).

DETAILED DESCRIPTION:
Previous studies showed that anodal transcranial direct current stimulation (atDCS) can have beneficial effects on word-retrieval in healthy younger and older subjects. The present study aims to extend these findings by assessing whether atDCS can also improve known impairments of word-retrieval in Mild Cognitive Impairment. atDCS will be applied to the left inferior frontal gyrus in a sham controlled cross-over within subjects design. Simultaneous functional magnetic resonance imaging (fMRI) will assess underlying neural effects of the stimulation.

ELIGIBILITY:
Inclusion Criteria:

* right handed
* German native speakers
* clinical diagnosis of Mild Cognitive Impairment

Exclusion Criteria:

* dementia
* other current or previous neurological or current psychiatric diseases
* alcohol or drug abuse
* MRI contraindication (e.g., magnetic metal, pacemaker, claustrophobia

Ages: 45 Years to 86 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2012-12; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Number of correct responses during word-generation tasks (max. 60) | Change in number of correct responses between Assessment 1 (week 1) and Assessment 2 (week 2), assessments 1 and 2 are seperated by one week
  Subjects are assessed in a cross-over design. The primary outcome measure will be assessed twice in each subject, either during sham stimulation or active stimulation with transcranial direct current stimulation. Order of stimulation (sham, atDCS or atDCS, sham) will be counterbalanced across the group. The study design has been described in detail before (Meinzer et al., 2012, Journal of Neuroscience, 32:1859 -1866).

SECONDARY OUTCOMES:
Neural activity during word-generation task assessed by functional magnetic resonance imaging (fMRI) | Change in fMRI activity between Assessment 1 (week 1) and Assessment 2 (week 2), assessments 1 and 2 are seperated by one week

CONTACTS AND LOCATIONS:
Overall Officials: Agnes Flöel, MD, Principal Investigator — Charite University Medicine, Department of Neurology
Locations (1):
- Charite University Medicine, Department of Neurology, Berlin, State of Berlin, Germany